CLINICAL TRIAL: NCT01632267
Title: A Retrospective Analysis of Outcomes in Outpatients With Major Depressive Disorder (MDD) in a Staff Model HMO: Pharmacogenetic Algorithm for Psychotropic Pharmacotherapeutic Applications
Brief Title: Retrospective Analysis of Outcomes With a Pharmacogenomic Algorithm
Acronym: UHS
Status: Completed | Type: Observational
Sponsor: Assurex Health Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 10003
Record Dates: First submitted 2012-06-27; First posted 2012-07-02 (Estimated); Results first posted 2013-03-22 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2013-02

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Buccal samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Depression and anxiety: Subjects with a primary diagnosis of depression or anxiety disorder.

SUMMARY:
Antidepressants are among the most widely prescribed medications, yet only 35-45% of patients achieve remission following an initial antidepressant trial. The financial burden of treatment failures in direct treatment costs, disability, decreased productivity, and missed work may in part derive from a mismatch between optimal, and actual, medications prescribed. The present one year retrospective study seeks to evaluate the indirect and direct healthcare costs for 96 patients with a DSM-IV-TR depressive or anxiety disorder, in relation to an interpretive reporting system designed to predict antidepressant responses based on DNA variations in cytochrome P450 genes (CYP2D6, CYP2C19, CYP1A2), the serotonin transporter gene (SLC6A4), and the serotonin 2A receptor (5HTR2A) genes.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder
* Dysthymic Disorder
* Depressive Disorder NOS
* Obsessive Compulsive Disorder (OCD)
* Generalized Anxiety Disorder
* Panic Disorder
* Anxiety Disorder NOS
* Post-Traumatic Stress Disorder (PTSD)
* Social Phobia

Exclusion Criteria:

* Bipolar Disorder
* Schizophrenia
* Schizoaffective Disorder
* Previous pharmacogenomic testing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects under the care of a psychiatrist at Union Health Services, Chicago, IL
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aida Spahic-Mihajlovic, MD, Principal Investigator — Union Health Services
Locations (1):
- Union Health Services, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Depression and Anxiety
Started | 104
Completed | 97
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Depression and Anxiety
Number analyzed (Participants) | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 97
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 104

OUTCOME MEASURES:

1. Primary Outcome: Number of Outpatient Visits
Description: Number of outpatient healthcare visits during study window
Time Frame: During the one year study window (April 1, 2010 to April 1, 2011)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depression and Anxiety
Number analyzed (Participants) | 97
units on a scale | 13 (9.4)

2. Secondary Outcome: Number of Medical Absence Days
Description: Number of medical absence days during study window
Time Frame: During the one year study window (April 1, 2010 to April 1, 2011)
Reporting Status: Not Posted

3. Secondary Outcome: Number of Disability Claims
Description: Number of disabiity claims during study window
Time Frame: During the one year study window (April 1, 2010 to April 1, 2011)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Depression and Anxiety
Serious Adverse Events (participants affected / at risk) | 0/104
Other Adverse Events (participants affected / at risk) | 0/104

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No